CLINICAL TRIAL: NCT04248491
Title: A Single-Blind, Randomized Study of the BTL Emsella Chair Versus Sham for the Treatment of Chronic Pelvic Pain
Brief Title: Emsella Chair Versus Sham for the Treatment of Chronic Pelvic Pain
Acronym: EmsellaPain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment and lack of efficiency
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-348
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Pain
Keywords: Chronic Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Patients who meet all the eligibility criteria will be enrolled in the study and randomized (1:1) to receive Emsella chair or sham treatments. The subject and biostatistician will be blinded to the group allocation throughout the study. The initial analysis of data, performed by the biostatistician will not include group assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The sham Emsella treatment will provide sensation without active HIFEM technology. The sham treatment amplitude setting will be limited to below the therapeutic level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Emsella Chair Active Treatment (Active Comparator): Subjects will be asked to sit on the device and the height will be adjusted until the subject's feet are on the floor. The active treatments are individualized, since some subjects will be more sensitive than others. The Emsella Chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will be decreased slightly and stay unchanged for the remainder of the treatment. The treatment threshold should be increased with every treatment until the subject reaches 100%.
  Interventions: Device: BTL Emsella chair
- Emsella Sham Treatment (Sham Comparator): Sham treatment subjects will be positioned on the device in the same manner. The sham treatment will provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below the therapeutic level (<10% power).
  Interventions: Device: BTL Emsella chair

INTERVENTIONS:
Device: BTL Emsella chair — Subjects will sit on the device. The Research Nurse Coordinator (RNC) will turn the device on and increase the setting gradually until the patient reaches their sensory threshold. This is the maximum sensation the patient can tolerate. The treatment threshold should be increased with every treatment until the subject reaches 100%.

SUMMARY:
The purpose of this clinical trial is to compare the Emsella Chair therapy to Sham and to determine whether electromagnetic technology is effective in the treatment of chronic pelvic pain. Currently there are no other studies utilizing the Emsella Chair for the treatment of chronic pelvic pain. Eligible subjects will receive 2 treatments per week for a total of 4 weeks.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a common and often debilitating in both men and women. It occurs below the umbilicus and is severe enough to cause functional impairment or require treatment. The health care burden of CPP is substantial. First line treatments involve a multidisciplinary approach and include general relaxation and stress management, patient education, self-care and behavioral modification, and pain management. Second-line agents include physical therapy (avoiding kegel exercises), and oral and intravesical agents. More invasive options including neuromodulation.

The Emsella chair is currently approved as a treatment for stress urinary incontinence. Chronic pelvic pain patients may benefit from treatment. The Emsella chair generates electromagnetic stimulation which is able to penetrate deep into the pelvic floor muscles inducing stimulation and providing rehabilitation for weak pelvic floor muscles. The Emsella chair is a novel high-intensity focused electromagnetic (HIFEM) technology for the treatment of stress urinary incontinence (SUI), in addition to other pelvic floor related disorders. HIFEM technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercises over 28 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written, dated, informed consent prior to screening, and be likely to comply with study protocol, including independently complete study questionnaires and communicate with study personnel about adverse events (AEs) and other clinically important information.
2. Females and males, 18 to 80 years of age, at screening
3. Self-reported CPP defined as pelvic pain that is non-cyclical and of at least 6 months duration and refractory to other treatments
4. Subject agrees not to start any new treatment for CPP (medication or otherwise) during the treatment and follow-up periods.
5. Subject agrees to maintain a stable dose all current medications throughout the treatment and follow-up period

   For Females Only:
6. If of child-bearing age and female, agree to practice approved birth-control methods (oral contraceptives, condom barrier, injection, diaphragm or cervical cap, vaginal contraceptive ring, Intrauterine device (IUD), implantable contraceptive, surgical sterilization (bilateral tubal ligation), vasectomized partner(s))

Exclusion Criteria:

1. Pelvic floor physical therapy, including muscle training and/or electrostimulation, in a clinical setting within 30 days prior to screening.
2. Pelvic floor trigger point injections, pudendal nerve block, or bladder hydrodistention within 30 days prior to screening
3. Subject weighs more than 330 pounds
4. Current urinary tract infection (UTI). If a subject has a confirmed symptomatic UTI at screening, per the investigator's clinical judgment, they will be deferred from screening until treatment is completed, and may resume once symptoms have resolved.
5. Pulmonary insufficiency, defined as difficulty breathing and fatigue, especially during exercise; heartbeat (palpitations); swelling of the legs or feet; dizziness or fainting; and/or bluish discoloration of the nails and/or lips (cyanosis)
6. Subject is currently receiving treatment for a malignant tumor that would interfere with study participation.
7. Any condition that causes a lack of normal skin sensation to the pelvis, buttocks, and lower extremities
8. History of Hunner's lesion in the medical record
9. Major metal implants such as: metal plates, screws, joint replacements, implanted cardiac pacemakers, drug pumps, neurostimulators, electronic implants, copper intrauterine devices, defibrillators, and metal implants in the pelvic area. Patients with other metal implants will be evaluated by the investigator for inclusion in the study.
10. Subject has a piercing between the waist and knees and is not willing to remove it before each treatment
11. Subject has used the BTL EMSELLA device previously
12. Currently participating in an investigational study that may impact study results or previously received an investigational drug or treatment within 30 days of the Screening Visit
13. Current or history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation

    For Females Only:
14. Pregnant, or planning to become pregnant, at screening or anytime throughout the study period

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital-Royal Oak
Locations (1):
- Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Emsella Chair Active Treatment: Subjects will be asked to sit on the device and the height will be adjusted until the subject's feet are on the floor. The active treatments are individualized, since some subjects will be more sensitive than others. The Emsella Chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will be decreased slightly and stay unchanged for the remainder of the treatment. The treatment threshold should be increased with every treatment until the subject reaches 100%.
  BTL Emsella chair: Subjects will sit on the device. The RNC will turn the device on and increase the setting gradually until the patient reaches their sensory threshold. This is the maximum sensation the patient can tolerate. The treatment threshold should be increased with every treatment until the subject reaches 100%.
- Emsella Sham Treatment: Sham treatment subjects will be positioned on the device in the same manner. The sham treatment will provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below the therapeutic level (<10% power).
  BTL Emsella chair: Subjects will sit on the device. The RNC will turn the device on and increase the setting gradually until the patient reaches their sensory threshold. This is the maximum sensation the patient can tolerate. The treatment threshold should be increased with every treatment until the subject reaches 100%.
Period: Overall Study
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 person in the active treatment group was lost to follow-up. Baseline demographic data was not available for this patient.
Groups:
- Total: Total of all reporting groups
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (17) | 36 (13) | 45 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 9
  American Indian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Change in Subject-reported Pain and Discomfort as Measured by the Visual Analog Scale (VAS)
Description: Mean change in Pain VAS from baseline to end of treatment will be compared between the Emsella Chair group and the sham group. VAS is scored from 0-10, where 0 = no pain and 10 = worst possible pain. Value at week 8 minus the value at baseline was used to calculate change. Negative numbers indicate an improvement in pain, and positive numbers indicate a worsening pain.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
units on scale | 0.6 (1.52) | 1.6 (1.82)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.342, t-test, 2 sided

2. Secondary Outcome: The Change in Subject-reported Impression of CPP Severity as Measured by the Patient Global Impression of Severity Scale (PGI-S).
Description: Change in subject-reported impression of CPP severity as measured by the Patient Global Impression of Severity scale (PGI-S). The subject will check the box that describes how their condition is now. This is a four point scale, with 1=normal, 2= mild, 3=moderate, and 4= severe. The value at week 12 minus the value at baseline was calculated. A positive change indicates a worsening condition, and a negative value indicated an improvement in condition.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
units on a scale | 0.2 (0.45) | -0.6 (0.55)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.035, t-test, 2 sided

3. Secondary Outcome: The Number of Participants Reporting Significant Symptom Improvement as Measured by the Patient Global Impression of Improvement Scale (PGI-I)
Description: Subject-reported impression of CPP improvement as measured by the Patient Global Impression of Improvement scale (PGI-I). The scale has 7 points with a lower number indicating improvement: (1=very much better, 2=much better, 3=a little better, 4=no change, 5=a little worse, 6-=much worse, 7= very much worse) to describe their chronic pelvic pain symptoms now versus prior to study treatment. We will report the number of individuals reporting a score of 1 or 2, very much better or much better (significantly improved).
Time Frame: at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

4. Secondary Outcome: The Change in Subject-reported Impression of CPP Severity as Measured by Subject-reported Pelvic Floor Tenderness to Palpation During 4 Quadrant Pelvic Examination as Measured by VAS.
Description: A trained provider will complete a pelvic (women) or rectal (men) exam on subjects. The VAS is a validated questionnaire that assesses pain on a scale from 0 = no pain to 10 = worst possible pain. The subject will provide a pain score from 0 - 10 for each of the 4 quadrants assessed. The average pain score of the 4 quadrants is then calculated. The average pain score ranges from 0 to 10. The value from baseline to secondary endpoint at week 12 is calculated. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
units on a scale | -0.05 (1.39) | 1.45 (1.14)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.098, t-test, 2 sided

5. Secondary Outcome: The Change in Subject-reported Impression of CPP Severity in Females.
Description: The change in CPP severity as measured by subject-reported sexual function as measured by the Female Sexual Function Index questionnaire (FSFI) for female subjects. The FSFI is a 19 question survey. A lower score is equivalent to a higher degree of sexual dysfunction. Scores range from 0 to 36. The change value is calculated from baseline to week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and Week 12
Population: 4 females were enrolled in the study. One was randomized to active treatment, 3 were randomized to sham treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 1 | 3
score on a scale | -2.20 (0) | 0.37 (2.21)

6. Secondary Outcome: The Change in Subject-reported Impression of CPP Severity in Males.
Description: The change in CPP severity as measured by subject-reported sexual function as measured by the Brief Sexual Function Inventory questionnaire (BSFI) for male subjects. The BSFI is a validated questionnaire for male sexual function. Average score ranges from 0 to 44. A lower score indicates a higher degree of dysfunction. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms. Calculated from the value at week 12 minus value at baseline
Time Frame: Baseline and week 12
Population: A total of 6 males were enrolled in the study. 4 were randomized to active treatment, 2 were randomized to sham treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 4 | 2
score on a scale | 0.575 (0.46) | -0.10 (0.14)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.192, t-test, 2 sided

7. Secondary Outcome: The Change in Subject-reported Depression Severity as Measured by the Beck Depression Inventory (BDI).
Description: The Beck Depression Inventory is a 21-question multiple-choice self-report inventory. It is composed of items relating to symptoms of depression such as hopelessness, irritability, guilt, fatigue, weight loss, and lack of interest in sex. Subjects that score greater than 30 at any time may be referred for psychological evaluation but may continue study participation. A higher score indicates a greater severity of depression. Scores can range from 0 to 63. The value of change calculated from baseline minus week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | -3.6 (7.5) | 3.0 (5.74)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.157, t-test, 2 sided

8. Secondary Outcome: The Change in Subject-reported Bother Related to Overactive Bladder Symptoms as Measured by the Overactive Bladder Questionnaire-Short Form (OAB-Q).
Description: Since both overactive bladder (OAB) and interstitial cystitis/bladder pain syndrome (IC/BPS) share urinary urgency and frequency symptoms, this validated measure will evaluate additional aspects associated with OAB and IC/BPS. The OAB-Q Short Form (SF) consists of two scales assessing symptom bother and health-related quality of life (HR-QOL) in patients with OAB. Each question is rated on a 6 point scale with 1 = Not at all and 6 = A very great deal. Scores can range from 0 to 100. The change value is calculated from the baseline value minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | 7.33 (10.38) | 7.33 (10.90)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 1.00, t-test, 2 sided

9. Secondary Outcome: The Change in Subject-reported Urinary and Pain Symptoms, as Well as Bother, as Measured by the Interstitial Cystitis Symptom Index and Problem Index (ICSI-PI).
Description: IC/BPS patients can share urinary urgency and frequency symptoms. The ICSI-PI measures urinary and pain symptoms and assesses how problematic are. A higher score indicates greater severity of symptoms. Scores range from 0-36. The change is calculated by the baseline value minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | 2.2 (1.79) | 1.2 (2.28)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.463, t-test, 2 sided

10. Secondary Outcome: The Change in Subject-reported Anxiety Symptoms as Measured by the Generalized Anxiety Disorder Questionnaire (GAD-7).
Description: The GAD-7 questionnaire is a 7-item validated scale to assess generalized anxiety disorder. Patients are grouped by GAD score 0-7 and 8+ which suggests no anxiety disorder and probably anxiety disorder, respectively. Scores can range from 0 to 21. The change is calculated as the value at baseline minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | -1.2 (4.76) | -1.8 (1.79)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.799, t-test, 2 sided

11. Secondary Outcome: The Change in Subject-reported Pain as Measured by the McGill Pain Questionnaire (MPQ).
Description: The McGill Pain Questionnaire can be used to evaluate a person experiencing pain over time to determine the effectiveness of an intervention. The questionnaire consists of 22 questions. Each question is scored 0 (none) to 10 (worst possible). A higher score indicates more severe pain symptoms. Scores range from 0 to 220. The change calculated from the value at baseline minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | 8.8 (22.11) | 5.2 (12.07)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.757, t-test, 2 sided

12. Secondary Outcome: The Change in Subject-reported Rumination, Magnification, and Helplessness Related to Pain as Measured by the Pain Catastrophizing Scale (PCS).
Description: The Pain Catastrophizing Scale (PCS) lists thirteen statements describing different thoughts and feelings that may be associated with pain. Each statement is rated as: 0 =not at all, 1= to a slight degree, 2= to a moderate degree, 3= to a great degree, and 4= all the time. Subjects who report a larger number associated with such thoughts during pain are more likely to rate the pain as more intense. Scores range from 0 to 52. The change is calculated as the value at baseline minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | 3.6 (11.06) | -0.6 (5.68)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.472, t-test, 2 sided

13. Secondary Outcome: The Subject-reported Perception of Overall Improvement in Pain as Measured by Global Response Assessments (GRA) for Pain and Quality of Life.
Description: The GRA is a 7-point scale to evaluate the subject's perception of overall improvement in pain. It is scored as follows: 1 = markedly worse, 2 = moderately worse, 3 = mildly worse, 4 = same (unchanged), 5 = slightly improved, 6 = moderately improved, and 7 = markedly improved. The number of participants reporting significant improvement in pain (score of 6 or 7) at week 12 are counted.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
Participants | 1 | 1

14. Secondary Outcome: Change in Subject-reported Pain and Discomfort as Measured by VAS
Description: Change in subject reported pain and discomfort as measured by the Visual Analog Scale (VAS). The VAS is a validated questionnaire that assesses pain on a scale from 0= no pain to 10= worst possible pain. The change is calculated from the value at baseline minus the value at week 12. Positive change indicates improvement of symptoms. A negative change indicates worsening of symptoms.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
score on a scale | -0.2 (0.84) | 0.8 (2.05)
Statistical Analysis 1: Comparison: Emsella Chair Active Treatment vs Emsella Sham Treatment; Test type: Superiority; p = 0.342, t-test, 2 sided

15. Secondary Outcome: Safety and Tolerability Will be Assessed as the Number of Esmella Chair-related With Adverse Events.
Description: Safety and tolerability of the Emsella chair compared to Sham will be assessed as the number of adverse events reported that were determined to be related to the Emsella chair treatment.
Time Frame: From baseline to week 12
Measure: Number; unit: Adverse events
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
Number analyzed (Participants) | 5 | 5
Adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Emsella Chair Active Treatment | Emsella Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emsella Chair Active Treatment (N=5) | Emsella Sham Treatment (N=5)
Covid infection (Infections and infestations) | 0 (0) | 2 (2)
Vaginal yeast infection (Infections and infestations) | 0 (0) | 1 (1)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Injury unrelated to procedure

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of efficacy at an interim analysis point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT04248491/Prot_SAP_000.pdf